CLINICAL TRIAL: NCT00857363
Title: SmartPill Colonic Transit Time Validation Study in Patients With Chronic Constipation
Brief Title: Colonic Transit Time Validation Study
Acronym: CTT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The SmartPill Corporation (Industry)
Responsible Party: Jack Semler/Chief Technology Officer, The SmartPill Corporation
Other Study IDs: 120508
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Constipation
Keywords: capsule; constipation; whole gut transit; colonic transit; gastric emptying; small bowel transit
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Constipated: Adult subjects with functional constipation as define by Rome II criteria

SUMMARY:
The protocol described herein is designed to provide clinical evidence of the substantial equivalence of SmartPill GI Monitoring System (SP) to the Sitzmarks (Konsyl Pharmaceuticals, Easton, MD) radio-opaque markers (ROM). The trial will enroll symptomatic subjects who meet Rome III criteria (1) for chronic functional constipation.

DETAILED DESCRIPTION:
The primary aim of this study is to assess the equivalence of SP to ROM through characterization of device agreement using SP cutoffs for colonic and whole gut transit (59hrs and 73 hrs respectively) derived from the above mentioned study. The cutoffs are derived from the 95th percentile of the healthy subjects in the study. Demonstration of agreement will also serve to validate these SP cutoffs. Device agreement will be evaluated by comparing the percentage of subjects identified with slow transit versus normal transit with SmartPill to the percentage of subjects identified with slow versus normal transit with ROM in the study population. The colonic transit time results will serve as the primary measure for slow versus normal transit for SmartPill. For ROM test we will employ the Metcalf protocol which provides a measure of whole gut transit to compare the SmartPill results to. Additionally, we will characterize gastric emptying and small bowel transit time of the SmartPill in this population. The SmartPill test will be administered simultaneously with ROM. A modified Metcalf procedure will be employed for characterization of slow transit by ROM.

The SmartPill GI Monitoring System offers an alternative non-invasive method for characterizing disorders of the stomach. The system consists of an ingestible capsule that houses sensors for pH, temperature, and pressure, a receiver for receiving and storing signals from the capsule, and software for displaying data on a personal computer. The capsule samples at regular intervals and transmits the sensed pH, pressure, and temperature data to a portable receiver worn by the subject. After test completion, the recorded data is downloaded to a personal computer for subsequent evaluation. This trial is for subjects 18 years of age to 80 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between ages of 18-80 years of age with symptoms of chronic functional constipation for at least one year.
2. Self reported bowel movement frequency of < 2 bowel movements/week for at least 3 of the last 6 months.
3. Presenting at least one of the following symptoms as defined by Rome III criteria

   * Feeling of incomplete evacuation with > 25% of bowel movements
   * Digital maneuvers with > 25% of bowel movements
   * Hard stools with > 25% of bowel movements
   * Feeling of blockage with > 25% of bowel movements
   * Straining with > 25% of bowel movements
4. Constipation, not abdominal pain, as the predominant symptom.
5. Ability to stop laxatives, prokinetic agents, and narcotic analgesic agents 3 days prior to SP and ROM ingestion visit and during the study period.
6. Ability to stop proton pump inhibitors for seven days and Histamine2 blockers for three days prior to and the day of SmartPill ingestion.
7. No evidence of metabolic disease (hypothyroidism, uncontrolled diabetes, electrolyte imbalance).
8. A normal colonoscopy or barium enema within 5 years for individuals over 50 years of age.

   -

Exclusion Criteria:

1. Participation in the previous SmartPill Whole gut transit Study titled "Assessment of Whole Gut Transit Time Using the SmartPill Capsule: A Multicenter Study" Protocol Number 122205
2. Previous history of bezoars.
3. Prior GI surgery except for cholecystectomy, appendectomy, or Nissen fundoplication
4. Any abdominal surgery within the past 3 months
5. Known or history of inflammatory bowel disease
6. History of diverticulitis, diverticular stricture, and other intestinal strictures
7. Tobacco use within eight hours prior to capsule ingestion and during the initial 8 hour recording on Day 0 or the Ingestion visit.
8. Alcohol use within eight hours prior to capsule ingestion and throughout the entire monitoring period (5 days).
9. BMI > 40 kg/m2
10. Allergies to components of the SmartBar (Appendix IX).
11. Females of childbearing age who are not practicing birth control and/or are pregnant or lactating. (A urine pregnancy test will be performed on female subjects prior to capsule ingestion). Acceptable forms of birth control include oral contraceptives, double barrier method, and IUD cover and must be practiced from the time of enrollment until the time of release from the study.
12. Cardiovascular, endocrine, renal, or other chronic disease likely to affect motility.
13. Use of medical devices such as pacemakers, infusion pumps, or insulin pumps.
14. Any contraindication to use of Fleets Enema.
15. Uncontrolled diabetes with a hemoglobin A1C greater than 10%.
16. Severe dysphagia to food or pills

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with constipation referred to a tertiary motility center
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-05 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Colonic Transit Time | 4 days and 7 days

SECONDARY OUTCOMES:
Determine regional gut (gastric, small bowel, colonic) transit times | continuous time measure until caspule elimination

CONTACTS AND LOCATIONS:
Overall Officials: John R Semler, PHD, Study Chair — The SmartPill Corporation
Locations (13):
- United States (12):
  - University of Arizona Health and Sciences Ctr Southern Arizona VA HealthCare System, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Med Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Med Center, Ann Arbor, Michigan
  - Jasper Clinic, Inc., Kalamazoo, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Buffalo VA Medical Center, Buffalo, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Wake Forest University Medical Center, Winston-Salem, North Carolina
  - Temple University Medical Center, Philadelphia, Pennsylvania
- Queen Mary, University of London, London, United Kingdom

REFERENCES:
- [Derived] Camilleri M, Thorne NK, Ringel Y, Hasler WL, Kuo B, Esfandyari T, Gupta A, Scott SM, McCallum RW, Parkman HP, Soffer E, Wilding GE, Semler JR, Rao SS. Wireless pH-motility capsule for colonic transit: prospective comparison with radiopaque markers in chronic constipation. Neurogastroenterol Motil. 2010 Aug;22(8):874-82, e233. doi: 10.1111/j.1365-2982.2010.01517.x. Epub 2010 May 11. PMID 20465593